CLINICAL TRIAL: NCT07261085
Title: A Real-world Study on the Effectiveness of Nirmatrelvir-ritonavir in Reducing Severe Outcomes From COVID-19
Brief Title: A Study to Learn How Paxlovid [Nirmatrelvir-ritonavir/PF-07321332] Works in COVID-19 Patients Who Are Elderly or Have Medical Conditions.
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4671071
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: COVID-19
Keywords: Covid-19; SARS-COV2
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Assessed and Treated Cohort: Participants who were assessed with Covid prescribed and subsequently dispensed nirmatrelvir-ritonavir during the selection period
  Interventions: Drug: nirmatrelvir-ritonavir
- Assessed and Untreated Cohort: Participants who were assessed with Covid for nirmatrelvir-ritonavir but either were not prescribed the medication or did not have it dispensed during the selection period
  Interventions: Other: No treatment

INTERVENTIONS:
Drug: nirmatrelvir-ritonavir — Participants who were assessed with Covid prescribed and subsequently dispensed nirmatrelvir-ritonavir during the selection period
  Other Names: paxlovid
  Groups: Assessed and Treated Cohort
Other: No treatment — Participants who were assessed with Covid for nirmatrelvir-ritonavir but either were not prescribed the medication or did not have it dispensed during the selection period
  Groups: Assessed and Untreated Cohort

SUMMARY:
The purpose of this study is to learn about the effects of the study medicine called Paxlovid [nirmatrelvir-ritonavir/PF-07321332], for the potential treatment of COVID-19.

This study will use patient health records in Ontario, to find people who were sick with COVID-19 and visited a pharmacist to be treated, anytime from December 1st, 2022, to March 31st, 2024. To be included in our study, the people must be over 18 years of age and be registered in the Ontario health system for at least one year. People were not included in our study if they have been pregnant in the past year or have serious kidney or liver disease.

We will separate the people in the study into two groups: those who received treatment with Paxlovid [nirmatrelvir-ritonavir/PF-07321332] and those who received no treatment. We will monitor their healthcare visits or if they die for any reason, for up to 60 days after the date that they visited their pharmacist. Then we will compare participant experiences when they are taking the study medicine to when they are not. This will help us determine if the study medicine is effective.

ELIGIBILITY:
Inclusion

* Record of at least 1 nirmatrelvir-ritonavir prescription and at least 1 dispensation issued by the pharmacist (Treated Cohort only) within 5 days of prescription, identified through pharmacy billing codes
* Record of at least 1 assessment for nirmatrelvir-ritonavir, without a prescription issued by the pharmacist (Untreated Cohort only), OR record of at least 1 prescription for nirmatrelvir-ritonavir without dispensation (Untreated Cohort only), identified through pharmacy billing codes

Exclusion

* Invalid or incomplete records (e.g., missing age, missing sex, death before index)
* Record of a positive PCR test for SARS-CoV-2 between 5 and 90 days prior to the index date
* Had a prescription for antivirals within 3 days prior to or on the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Institute for Clinical Evaluative Sciences (ICES) data repository consists of de-identified, record-level, coded and linkable health data sets. It encompasses much of the publicly funded administrative health services records for the Ontario population eligible for universal health coverage since 1986 and integrates administrative data, registries, and surveys.
Sampling Method: Non-Probability Sample
Enrollment: 99000 (Actual)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Time to the first severe composite outcome (all-cause hospital admission, ICU admission, or death) within 30 days of treatment assessment. | Participants selected between 01 Dec, 2022 to 31 March 2024

SECONDARY OUTCOMES:
Time to the first severe composite outcome (all-cause hospital admission, ICU admission, or death) within 60 days of treatment assessment. | Participants selected between 01 Dec, 2022 to 31 March 2024

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671071